CLINICAL TRIAL: NCT02559869
Title: Imaging and BioFluid Biomarkers in Amyotrophic Lateral Sclerosis
Acronym: TRACK-ALS
Status: Completed | Type: Observational
Sponsor: Massachusetts General Hospital (Other)
Collaborators: The Methodist Hospital Research Institute (Other); Cedars-Sinai Medical Center (Other); ALS Association (Other)
Responsible Party: Principal Investigator, Suma Babu, Co-Principal Investigator, Massachusetts General Hospital
Other Study IDs: 2015P000140
Record Dates: First submitted 2015-09-23; First posted 2015-09-24 (Estimated); Last update posted 2020-05-21 (Actual); Status verified 2020-05

CONDITIONS: Amyotrophic Lateral Sclerosis (ALS)
Keywords: Biofluid; ALS; MRI; PET; Imaging; Biomarkers; Amyotrophic Lateral Sclerosis; TRACK ALS; pathology
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis | interventions — GE-180; Ligands

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — iPSC Line Generation, DNA, Inflammatory Markers, Plasma, CSF
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Amyotrophic Lateral Sclerosis (ALS): Subjects will be diagnosed with possible, probable, probable-lab supported, or definite ALS.
  Interventions: Drug: [18F] GE-180
- Healthy Controls: Subjects with no known neurological disorder.
  Interventions: Drug: [18F] GE-180

INTERVENTIONS:
Drug: [18F] GE-180 — PET Tracer Ligand
  Other Names: ligand; PET Tracer

SUMMARY:
This is a multicenter, 18-month study, which aims to identify imaging and biofluid biomarkers in people with ALS to expand the understanding of ALS pathology, treatment targets, disease progression, and anatomical differences between different disease phenotypes. This pilot project is tailored to produce imaging tools that will allow researchers to conduct future ALS clinical trials more efficiently which may in turn impact the pace for ALS drug discovery.

DETAILED DESCRIPTION:
In this trial, approximately 200 subjects will participate in this study from 2 Northeast ALS Consortium (NEALS) centers in the United States. Fifty (50) ALS participants will be age and gender matched to 50 participants with no known neurological disorder (healthy controls). Of these, twenty five (25) ALS participants will be age (±5 years) gender and binding affinity (TSPO) matched to 25 healthy controls.

During the enrollment period 200 participants will be screened and 100 participants will ultimately be scanned. There will be a maximum allowed time of 45 days between the screening and baseline visits (1st scan). All 100 subjects will undergo MRI scanning and clinical assessment at the Baseline Visit. Healthy control participants will have no further follow-up visits once they have completed their participation in the screening and baseline visits. Only 50 subjects from this sample will undergo PET scanning. The ALS participants will return for follow-up MRI scanning and clinical assessments every three months and follow-up PET scanning every 6 months over a 12-month period.

ELIGIBILITY:
Inclusion Criteria

Study subjects meeting all of the following criteria will be allowed to enroll in the study:

1. Male or female, aged 18 to 80
2. Medically safe to undergo MRI scans
3. Able to safely lie supine for at least 90 minutes in the opinion of the Site Investigator
4. Capable of providing informed consent and following trial procedures
5. Geographically accessible to the site

ALS subjects must also meet the following criteria:

1. Sporadic or familial ALS diagnosed as possible, laboratory-supported probable, probable, or definite as defined by modified El Escorial criteria
2. ALS Cognitive Behavioral Screen score >10 on the cognitive scale and/or >32 on the behavioral scale

Those ALS subjects participating in the optional lumbar puncture portion of the study must also meet the following criteria:

1. Subjects medically able to undergo lumbar puncture (LP) as determined by the investigator (i.e., no bleeding disorder, allergy to local anesthetics, a skin infection at or near the LP site, or evidence of high intracranial pressure).

For those subjects participating in the PET scan portion of the study, subjects must also meet the following criteria:

1. Medically safe to undergo PET scans
2. No prior radiation exposure that exceeds the site's current guidelines
3. No known allergy to any components of the tracer
4. Baseline ECG values are within normal range
5. Subjects must meet main study entry criteria

Exclusion Criteria

Study subjects meeting any of the following criteria during screening evaluations will be excluded from entry into the study:

1. Any contraindication to undergo MRI studies such as

   1. History of a cardiac pacemaker or pacemaker wires
   2. Metallic particles in the body
   3. Vascular clips in the head
   4. Prosthetic heart valves
   5. Claustrophobia
2. Diagnosis of Parkinson's disease or Alzheimer's disease
3. Diagnosis of renal failure
4. Have active or chronic autoimmune disease (such as hepatitis or HIV), infection, or taking immunosuppressive medications such as steroids, cyclophosphamide, etc.
5. Presence of diaphragm pacing system (DPS)
6. The presence of unstable psychiatric disease, cognitive impairment, or dementia that would impair ability of the subject to provide informed consent, according to SI judgment
7. Pregnant women or women currently breastfeeding
8. Anything that, in the opinion of the investigator, would place the subject at increased risk or preclude the subject's full compliance with or completion of the study

In addition, any subject meeting any of the following criteria during screening evaluations will be excluded from entry into the PET portion of the study:

1. Radiation exposure that exceeds the site's current guidelines
2. Low affinity TSPO binders determined by having a Thr/Thr polymorphism in the TSPO gene (rs6971) at the Screening Visit

Women of Childbearing Potential (WOCBP) For the purposes of this study, women of child bearing potential are defined as all women who are capable of becoming pregnant, unless they meet one of the following criteria:

* 12-months post-menopausal
* Post-hysterectomy
* Surgically sterile

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Approximately 200 subjects will be screened and approximately 100 subjects will be enrolled. Fifty (50) subjects will be diagnosed with possible, probable, probable-lab supported, or definite ALS, fifty (50) subjects will have no known neurological disease.
Sampling Method: Non-Probability Sample
Enrollment: 86 (Actual)
Dates: Start 2015-11; Primary Completion 2019-06-28 (Actual); Study Completion 2019-06-28 (Actual)

PRIMARY OUTCOMES:
Measure & localize brain inflammation in people with ALS via [18F] GE-180 PET imaging. | 12 months
  Aim 1 will be accomplished by obtaining [18F] GE-180 PET imaging from 25 people with ALS compared to 25 age, gender, and binding affinity matched healthy volunteers.
Define anatomical, structural, and functional changes in the brain via MRI of ALS Subjects vs. Healthy Controls at Baseline | 12 months
  Aim 1 will be accomplished by obtaining state of-the-art MRI acquisition sequences from 50 people with ALS compared to 50 MRI age- and gender-matched healthy volunteers.
Determine systemic inflammatory factors that may modify the progression or other clinical or imaging correlates of ALS. | 12 months
  Blood from 100 subjects will be studied to quantitate circulating pro- and anti-inflammatory monocyte/macrophage and T cells, with results to be correlated with neuroimaging and evaluated as potential biomarkers of disease progression.

SECONDARY OUTCOMES:
Determine the longitudinal changes in brain inflammation in people with ALS in correlation with ALS severity and rate of progression. | 12 months
  Clinical and [18F] GE-180 PET imaging data will be collected every 6 months from the 25 people with ALS for at least 12 months.
Determine the longitudinal changes in the anatomical, structural, and functional measures in people with ALS, and build ALS prediction models using the clinical and MRI data. | 12 months
  Clinical and MRI data will be collected every 3 months from 50 people with ALS for at least 12 months.

CONTACTS AND LOCATIONS:
Overall Officials: Suma Babu, MD, Principal Investigator — Massachusetts General Hospital; Joseph Masdeu, MD, PhD, Principal Investigator — Houston Methodist Neurological Institute
Locations (2):
- United States (2):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Houston Methodist Hospital, Houston, Texas

REFERENCES:
- See also: NEALS website (Northeast ALS Consortium) — http://alsconsortium.org